CLINICAL TRIAL: NCT06747572
Title: A Study to Determine the Prevalence and Clinical Characteristics Associated With PKD1 Gene Variant Groups in Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Brief Title: Polycystic Kidney Disease 1 (PKD1) Gene Variant Groups in Autosomal Dominant Polycystic Kidney Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: VX24-KDO-901; NL88429.078.24 (Registry Identifier: Overview of Medical Research in the Netherlands (OMON))
Record Dates: First submitted 2024-12-10; First posted 2024-12-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-12

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Keywords: ADPKD
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Part A: Eligible participants will complete a single visit to complete a blood sample collection for PKD1/2 genotyping.
- Part B: Participants who have completed all assessments in Part A and have a subset of variants in PKD1 will complete 1 year of follow-up.

SUMMARY:
The purpose of this study is to estimate the prevalence, demographic, and clinical characteristics of PKD1/2 gene variant groups in the ADPKD population.

ELIGIBILITY:
Key Inclusion Criteria:

* Estimated glomerular filtration rate (eGFR) greater than or equal to (≥) 30 milliliter per minute (mL/min)/1.73 m^2
* Willing and able to comply with scheduled visits and other study procedures
* A pre-existing diagnosis of ADPKD as defined in the protocol

Key Exclusion Criteria:

* History of kidney disease other than ADPKD that in the opinion of the investigator would independently impact the natural history of ADPKD
* History of solid organ or bone marrow transplantation or nephrectomy
* Ongoing renal replacement therapy or planning to start renal replacement therapy less than or equal to (≤)12 months from the Genotyping Visit in Part A

Other protocol defined Inclusion/Exclusion criteria will apply.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Part A: Male and female participants aged 12 to 65 years old, inclusive, diagnosed with ADPKD who have not reached end stage kidney disease (ESKD). Part B: Male and female participants aged 12 to 65 years old, inclusive, who have completed Part A and who have genotyping results confirming an eligible non-truncating variant in PKD1 and who are at risk for rapidly progressive disease, based upon historical total kidney volume (TKV) or kidney length.
Sampling Method: Non-Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Part A: Percentage of PKD1 Gene Variant Groups in the ADPKD Population | Genotyping Visit on Day 1 of Part A (Part A duration: 1 Calendar Day)
Part A: Weight of Participants Within Each PKD1 Gene Variant Group | Genotyping Visit on Day 1 of Part A (Part A duration: 1 Calendar Day)
Part A: Height of Participants Within Each PKD1 Gene Variant Group | Genotyping Visit on Day 1 of Part A (Part A duration: 1 Calendar Day)
Part A: Body Mass Index (BMI) of Participants Within Each PKD1 Gene Variant Group | Genotyping Visit on Day 1 of Part A (Part A duration: 1 Calendar Day)
Part A: Age of Participants at ADPKD Diagnosis Within Each PKD1 Gene Variant Group | Genotyping Visit on Day 1 of Part A (Part A duration: 1 Calendar Day)

CONTACTS AND LOCATIONS:
Locations (45):
- United States (27):
  - Alabama Kidney Research, Alabaster, Alabama
  - University of Alabama at Birmingham- Nephrology Research Clinic, Birmingham, Alabama
  - Kaiser Permanente - Los Angeles Medical Center, Los Angeles, California
  - UCLA Division of Nephrology, Los Angeles, California
  - Helen Diller Medical Center at Parnassus Heights, San Francisco, California
  - Nephrology & Hypertension Associates, PC, Middlebury, Connecticut
  - Yale Nephrology Clinical Research Clinic, New Haven, Connecticut
  - Nature Coast Clinical Research - Inverness, Inverness, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Emory School of Medicine - Renal Division, Atlanta, Georgia
  - Renal Associates, LLC, Columbus, Georgia
  - UChicago Medicine - Duchossois Center for Advanced Medicine - Nephrology, Chicago, Illinois
  - University of Iowa Health Care Medical Center- Nephrology, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - General Clinical Research Center, University of Maryland Baltimore, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center - Nephrology, Boston, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - University of Minnesota -Health Clinical Research Unit, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - DaVita Clinical Research, Las Vegas, Nevada
  - Columbia University Medical Center, New York, New York
  - Geisinger Clinic, Danville, Pennsylvania
  - Perelman Center for Advanced Medicine - Nephrology, Philadelphia, Pennsylvania
  - Nephrology Clinical Trials Center, Nashville, Tennessee
  - UVM Medical Center - 1 South Prospect Street, Burlington, Vermont
  - Swedish Center for Comprehensive Care, Seattle, Washington
- Belgium (2):
  - Universite Catholique de Louvain, Cliniques universitaires Saint-Luc (UCLouvain), Brussels
  - Universitaire Ziekenhuizen Leuven, Leuven
- Canada (2):
  - St. Joseph's Healthcare - Hamilton, Hamilton
  - MUHC - Montreal Children's Hospital, Montreal
- France (2):
  - Hopital de la Cavale Blanche, Brest
  - Necker Hospital, Paris
- Germany (2):
  - Charité - Klinik für Nephrologie und Intensivmedizin der, Berlin
  - Universitaetsklinik Koeln Department II of Internal Medicine, Cologne
- Netherlands (2):
  - UMCG - Nephrology, Groningen
  - Erasmus Medisch Centrum - Nephrology, Rotterdam
- FDI Clinical Research - San Juan, San Juan, Puerto Rico
- Hospital Fundacion Jimenez Diaz, Madrid, Spain
- United Kingdom (6):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - King's College Hospital, London
  - Royal Free NHS Trust, London
  - St Georges University Hospitals NHS Foundation Trust, London
  - Newcastle upon Tyne Hospitals NHS Foundation Trust - Freeman Hospital - Nephrology, Newcastle upon Tyne
  - Northern General Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/